CLINICAL TRIAL: NCT04387539
Title: A Sofosbuvir-based Quadruple Regimen is Highly Effective in HCV Type 4-infected Egyptian Patients With DAA Treatment Failure
Brief Title: ٍٍSofosbuvir/Simeprevir/Daclatasvir/Ribavirin and HCV Genotype 4-infected Egyptian Experienced Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOF/SMV/DCV/RBV
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Chronic HCV GT4; Sofosbuvir; Simeprevir; Daclatasvir; Ribavirin; Experienced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Cirrhotic (Active Comparator): SOF plus DCV/SMV/RBV regimen was administered to Egyptian non-cirrhotic experienced HCV GT4 participants for 12 weeks
  Interventions: Drug: SOF/SMV/DCV/RBV
- Cirrhotic (Active Comparator): SOF plus DCV/SMV/RBV regimen was administered to Egyptian cirrhotic experienced HCV GT4 participants for 12 weeks
  Interventions: Drug: SOF/SMV/DCV/RBV

INTERVENTIONS:
Drug: SOF/SMV/DCV/RBV — SOF was given orally at a dose of 400 mg/day DCV was given orally at a dose of 60 mg/day SMV was given orally at a dose of 150 mg/day. RBV was given in a total daily oral dose of 600 mg/day up to 1,200 mg/day according to the participant's weight and tolerability.
  Other Names: Olysio is a trade name of simeprevir; Sovaldi is a trade name of sofosbuvir; Daklinza is a trade name of daclatasvir

SUMMARY:
Experienced participants who had HCV GT4 infection were treated with Sofosbuvir/Simeprevir/Daclatasvir/Ribavirin (SOF/SMV/DCV/RBV)

DETAILED DESCRIPTION:
Experienced participants, who had chronic infection with HCV GT4 , and failed prior DAA treatments, SOF/DCV (71/92) or SOF/SMV (15/92) or SOF/pegylated interferon/RBV (2/92) or SOF/RBV (4/92) were enrolled in the current study.

In the present study, the regimen used was designed by the combination of triple DAAs with different mechanisms of action and non-overlapping resistance profiles, SOF/SMV/DCV, plus RBV.

ELIGIBILITY:
Inclusion Criteria:

* Experienced Egyptian participants with HCV GT4 infection who had failed prior DAA treatments [SOF/DCV or SOF/SMV or SOF/pegylated interferon/RBV or SOF/RBV]
* Fibrosis-4 score in non-cirrhotic participants is <1.45-3.25: (None or moderate fibrosis)
* Fibrosis-4 score in cirrhotic participants is >3.25: (Advanced fibrosis or cirrhosis)

Exclusion Criteria:

* HCV coinfected with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* had any liver disease other than chronic HCV GT4 infection.
* had a history of liver decompensation
* serum a-fetoprotein (AFP) > 100 ng/ml
* evidence of hepatocellular carcinoma
* major severe illness such as respiratory, renal, heart failure or autoimmune disease
* non-compliance with treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Each Treatment Arm | 12 weeks after last dose
  SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) level < 15 IU/m 12 weeks after the last dose of drugs.
Number of Participants With Adverse Events in Each Treatment Arm | Screening up to 12 weeks after last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a participant clinical investigation after administering a pharmaceutical drugs Serious adverse event (SAE) is an event that results in death, life-threatening, requires hospitalization, or significant disability/incapacity

SECONDARY OUTCOMES:
Percentage of Participants With Viral relapse | Up to 12 weeks after last dose
  Viral relapse was HCV RNA level undetectable at End of Treatment (EOT) (≤ 15 IU/ml), but detectable HCV RNA ( > 15 IU/ml) levels 12 weeks after planned EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdel-Gabbar, Ass. Prof, Principal Investigator — Biochemistry Dep., Faculty of Science, Beni-Suef University, P.O. Box 52621
Locations (1):
- Health Administration at Beni-Seuf, Bani Sweif, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Moneim A, Aboud A, Abdel-Gabbar M, Zanaty MI, Ramadan M. A sofosbuvir-based quadruple regimen is highly effective in HCV type 4-infected Egyptian patients with DAA treatment failure. J Hepatol. 2018 Jun;68(6):1313-1315. doi: 10.1016/j.jhep.2018.03.010. Epub 2018 Apr 3. No abstract available. PMID 29625827